CLINICAL TRIAL: NCT01138319
Title: Mitochondrial Mutations and AML
Brief Title: Biomarkers in Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B6; COG-AAML10B6 (Other: Children's Oncology Group); CDR0000671467 (Other: Clinical Trials.gov); NCI-2011-02224 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia; childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: DNA analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether clonally expanded somatic mitochondrial DNA mutations are associated with acute myeloid leukemia.

OUTLINE: Genomic DNA from blood samples obtained at diagnosis, remission, and relapse are analyzed for mitochondrial DNA mutations via PCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Available blood samples from diagnosis, remission, and relapse

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Association between clonally expanded somatic mitochondrial DNA mutations and acute myeloid leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Jason H. Bielas, PhD, Principal Investigator — Fred Hutchinson Cancer Center